CLINICAL TRIAL: NCT03291756
Title: CorEvitas Multiple Sclerosis (MS) Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: CorEvitas (Network)
Responsible Party: Sponsor
Other Study IDs: CorEvitas-MS-700
Record Dates: First submitted 2017-08-24; First posted 2017-09-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: Multiple Sclerosis Pts presenting to enrolling sites across the US are invited to enroll if eligible

SUMMARY:
This prospective, non-interventional research registry is designed to study the comparative effectiveness and comparative safety of approved treatments for MS in a cohort of patients cared for by neurologists across North America. Secondary objectives include analyzing the epidemiology and natural history of the disease, its comorbidities, and current treatment practices.

DETAILED DESCRIPTION:
The objective of the CorEvitas Multiple Sclerosis (MS) Registry is to create a national cohort of patients with MS. Data collected will be used to better characterize the natural history of the disease and to extensively evaluate the effectiveness and safety of medications approved for the treatment of MS. This will be done through the standardized collection of validated patient-reported outcomes (PRO) and clinician-reported outcomes (ClinRO), the prevalence and incidence of comorbidities and adverse events, medication utilization patterns and patient productivity measures.

The design is a prospective, non-interventional, observational registry for patients with MS under the care of a licensed neurologist. Longitudinal follow-up data is collected from both patients and their treating neurologist (also known as "Providers" for a CorEvitas registry study) every 6 months (+/- 30 days) during routine clinical encounters using CorEvitas registry forms. These forms collect data on patient demographics, disease duration, medical history (including all prior and current treatments for MS), smoking status, alcohol use, disease activity and severity, pain, as well as other clinician- and patient-reported outcomes, comorbidities and adverse events, infections, hospitalizations, and other targeted safety outcomes. After the enrollment visit, MS patients and physicians will complete the follow-up questionnaires during regularly scheduled clinical encounters. The goal is to collect data from patients and providers at six month intervals. Adverse events may be volunteered spontaneously by the subject, or be discovered as a result of general questioning by the Investigator. During all CorEvitas related visits with the Investigator, subjects will be questioned regarding the occurrence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of MS at the time of enrollment.
2. Age 18 years or older at the time of enrollment.
3. Willing to provide Personal Information.
4. Initiating (prescribed or starting) an Eligible Medication for the treatment of MS at the enrollment visit.

Exclusion Criteria:

1) Is participating or planning to participate in a double-blind randomized trial for an MS drug. Note: Concurrent participation in another observational registry or open-label Phase 3b/4 trial is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are enrolled in the Multiple Sclerosis (MS) Registry during regularly -scheduled office visits. Selected neurologists are invited to participate as investigators in the Registry.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-08-10 (Actual); Primary Completion 2100-12 (Estimated); Study Completion 2100-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events (AEs) or serious adverse events (SAEs). | Time Frame: A minimum of 10 years from last patient enrolled
  Targeted events include malignancy, anaphylaxis, cardiovascular disease, serious infection, autoimmune disease, MS Relapse, hepatic events, and general serious adverse events.
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

SECONDARY OUTCOMES:
Patient reported: Patient Clinical Global Impression (PCGI) Scale | Time Frame: every 6 months for 10 years
Disease burden: Relapse Information | Time Frame: every 6 months for 10 years
Percentage of patients with history of comorbidities | Time Frame: at registry enrollment
Physician reported: Nine-Hole Peg Test (9-HPT) | Time Frame: every 6 months for 10 years
Physician reported: Symbol Digit Modalities Test (SMDT) | Time Frame: every 6 months for 10 years
Patient reported: Patient reported: Work productivity and Activity Impairment (WPAI) | Time Frame: every 6 months for 10 years
Patient reported: Patient reported :MS Quality of Life, MSIS-29 | Time Frame: every 6 months for 10 years
Patient reported: MS Disability Score29 | Time Frame: every 6 months for 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- CorEvitas, LLC, Waltham, Massachusetts, United States

REFERENCES:
- See also: CorEvitas home page — https://www.corevitas.com/